CLINICAL TRIAL: NCT02879539
Title: Clinical Assessment of a Low Power Strategy for Cochlear Implant Recipients
Brief Title: Cochlear Implant Low Power Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Royal Victoria Eye and Ear Hospital (Other Government); Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC5607
Record Dates: First submitted 2016-08-21; First posted 2016-08-25 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: cochlear implants, power consumption,
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP3000-ACE strategy (Experimental): MP3000 sound coding strategy or ACE strategy with lower stimulation rate
  Interventions: Device: MP3000 sound coding strategy or ACE strategy with lower stimulation

INTERVENTIONS:
Device: MP3000 sound coding strategy or ACE strategy with lower stimulation

SUMMARY:
Reducing power consumption in the cochlear implant is crucial to the development of future smaller sound processors. The commercial MP3000 sound coding strategy has been shown to be more efficient in power consumption to the standard ACE strategy. However in order to develop smaller sound processors, further battery life power savings are required. The aim of this study is to evaluate three experimental sets of MP3000 parameter sets, compared against the default ACE program. In the background for each of the four strategies, experimental noise reduction programs (SpatialNR and NR3) will also be in use. In an additional phase of the study, low stimulation rate ACE programs will also be evaluated against the default stimulation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years) cochlear implant recipients
2. Implanted with the CI500, CI24RE and Nucleus 24 Series and CI422 cochlear implants.
3. User of commercially available Freedom, CP810 or CP900 series sound processor
4. User of the ACE strategy or MP3000 strategy
5. At least 3 months experience with the cochlear implant
6. Native speaker in the language used to assess speech perception performance
7. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Additional handicaps that would prevent participation in evaluations
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Word recognition scores in quiet | Testing over 18 weeks
  Word recognition scores in quiet for i) MP3000 strategy compared to default ACE strategy and ii) lower rate stimulation for ACE strategy
Sentence recognition scores in quiet | Testing over 18 weeks
  Sentence recognition scores in quiet for i) MP3000 strategy compared to ACE strategy and ii) lower rate stimulation for ACE strategy

SECONDARY OUTCOMES:
Fundamental frequency (F0) discrimination | Testing over 18 weeks
  F0 discrimination for MP3000 strategy compared to the ACE baseline
Speech intelligibility and helpfulness subjective ratings | Testing over 18 weeks
  For MP3000 strategy compared to the default ACE baseline
Sentence in noise scores | Testing over 18 weeks
  Comparison of MP3000 program with Spatial NR and NR3 enabled versus disabled.

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No